CLINICAL TRIAL: NCT01802307
Title: Focal Therapy for the Treatment of Organ Confined Prostate Cancer
Brief Title: Focal Therapy for Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00054478
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Focal therapy; Brachytherapy; Active surveillance; low risk cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Seeds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Focal Therapy (Experimental)
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Brachytherapy
  Other Names: Seeds

SUMMARY:
Prostate cancer is the most common solid organ cancer among men and is the second leading cause of cancer death. In 2013 about 238,590 men will be diagnosed with prostate cancer and 29,720 men will die of the cancer. Overall, about 1 in 6 men will be diagnosed with prostate cancer in their lifetime, but only 1 in 36 men will die. Currently, there are over 2.5 million men in the US living with prostate cancer. Standard treatment for prostate cancer has involved either removal of the prostate (radical prostatectomy) or application of some type of energy to the entire prostate gland in order to kill all of the cells--usually with radiation or cryotherapy (freezing).

Over the past decade, it has become apparent that while some men will benefit from treatment for prostate cancer, many will not. Particularly for men with a small amount of low-grade (not very aggressive) type of prostate cancer, the risk of death from this very slow-growing cancer is very low. However, the risk of harm from some of the treatments for prostate cancer is very high. Treatment for prostate cancer can cause erectile dysfunction, urinary leakage, difficulty urinating and overactive bladder and bowel symptoms.

One strategy for men with low risk prostate cancer has been to avoid immediate treatment and wait until the cancer starts to grow. The risk of this strategy is that some men may not be able to be cured once the cancer starts to grow. In addition, men who are on this active surveillance protocol can become very nervous, fearing that the cancer will start to spread.

A new strategy to avoid some of the treatment harms of prostate cancer while also attempting to avoid allowing the cancer to grow is called focal therapy. Many men with low-risk prostate cancer will have only a small piece of cancer within the prostate gland. These men may benefit from treating only this one area instead of the entire prostate. This will allow the physician to kill the cancer cells and to avoid some of the problems associated with treating the entire prostate.

The purpose of this study is to investigate the use of focal, targeted treatment of prostate cancer, that is, to treat only the small area of cancer instead of the entire prostate. We hope to show that this strategy will reduce the amount of side effects without compromising cancer cure.

DETAILED DESCRIPTION:
Prostate cancer is a lethal disease for ~11% of the men who are diagnosed with it. Early detection of prostate cancer using the PSA blood test can detect cancer a decade or more before it would have been found on a prostate examination. Men who are diagnosed at an older age (>75) may not benefit from aggressive treatment because many will not live long enough for the prostate cancer to kill them. Men who are diagnosed at a young age will be more likely to benefit from treatment from prostate cancer but they will have a very long time to live with some of the side effects of treatment.

Patients with low-risk prostate cancer, which is located in only one area or on one side of the prostate, may benefit from treatment of that one area instead of treating the entire prostate. This is similar to the lumpectomy of breast cancer which removes only the tumor instead of removing the entire breast.

This study will look at the short-term side-effects and the long-term success of performing focal treatment of prostate cancer.

Patients who are newly diagnosed with prostate cancer or who are already diagnosed and on an active surveillance protocol will be considered eligible for consideration of focal therapy. Patients deemed eligible will be offered inclusion in the study. There will only be a treatment group, no controls or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age >44
* Low risk Prostate Cancer (PSA <10, Gleason 6)
* Low-volume intermediate risk prostate cancer (PSA <15, Gleason 3+4=7)
* Organ confined disease

Exclusion Criteria:

* Metastatic Disease
* Palpable disease bilaterally
* Locally advanced disease either by digital rectal exam or MRI
* PSA >10 (for age <75)
* PSA >15

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Transrectal Ultrasound-guided prostate biopsy | yearly up to 5 years
  Annual prostate biopsy will determine oncological efficacy of treatment of the primary lesion. A standard 12 core biopsy will be performed with an additional 2 cores directed toward the area that was treated. Outcomes will be reported as 1) Presence/absence of cancer in the treated location and 2) Presence of new cancer lesions in other portions of the prostate.

SECONDARY OUTCOMES:
Erectile function | every 3-6 months for 5 years
  We will evaluate for any change from baseline and subsequent recovery of erectile function. Erectile function will be measured at baseline, then at 3-6 month intervals following treatment using a validated questionnaire, the International Index of Erectile Function (IIEF-5).
Urinary function/bother | every 3-6 months up to 5 years
  We will evaluate the change from baseline and degree of recovery of urinary function using a validated questionnaire, the International Prostate Symptom Score. Incontinence will also be assessed as present/absent and the number of pads used, if any.

CONTACTS AND LOCATIONS:
Overall Officials: James F Borin, MD, Principal Investigator — University of Maryland, College Park; Michael J Naslund, MD, Study Chair — University of Maryland, College Park
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Barret E, Ahallal Y, Sanchez-Salas R, Galiano M, Cosset JM, Validire P, Macek P, Durand M, Prapotnich D, Rozet F, Cathelineau X. Morbidity of focal therapy in the treatment of localized prostate cancer. Eur Urol. 2013 Apr;63(4):618-22. doi: 10.1016/j.eururo.2012.11.057. Epub 2012 Dec 13. PMID 23265382
- [Background] Klotz L. Active surveillance for prostate cancer: overview and update. Curr Treat Options Oncol. 2013 Mar;14(1):97-108. doi: 10.1007/s11864-012-0221-5. PMID 23318986
- [Background] Wilt TJ, Brawer MK, Jones KM, Barry MJ, Aronson WJ, Fox S, Gingrich JR, Wei JT, Gilhooly P, Grob BM, Nsouli I, Iyer P, Cartagena R, Snider G, Roehrborn C, Sharifi R, Blank W, Pandya P, Andriole GL, Culkin D, Wheeler T; Prostate Cancer Intervention versus Observation Trial (PIVOT) Study Group. Radical prostatectomy versus observation for localized prostate cancer. N Engl J Med. 2012 Jul 19;367(3):203-13. doi: 10.1056/NEJMoa1113162. PMID 22808955
- [Background] Suardi N, Capitanio U, Chun FK, Graefen M, Perrotte P, Schlomm T, Haese A, Huland H, Erbersdobler A, Montorsi F, Karakiewicz PI. Currently used criteria for active surveillance in men with low-risk prostate cancer: an analysis of pathologic features. Cancer. 2008 Oct 15;113(8):2068-72. doi: 10.1002/cncr.23827. PMID 18792067